CLINICAL TRIAL: NCT00083915
Title: University of Arkansas (UARK 2001-12), A Phase III Study of DTPACE Followed by Tandem Transplant With MEL 200 Versus MEL/DTPACE Hybrid and DTPACE Consolidation in Patients With Active Multiple Myeloma
Brief Title: DTPACE Followed by Tandem Transplant With Melphalan (MEL) 200 Versus MEL/Dexamethasone/Thalidomide (DT) Platinol/Adriamycin/Etoposide (PACE) Hybrid and DTPACE Consolidation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UARK 2001-12
Record Dates: First submitted 2004-06-03; First posted 2004-06-04 (Estimated); Results first posted 2011-08-03 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-10

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; DTPACE; Tandem Transplant; Cisplatin; Cyclophosphamide; Dexamethasone; Doxorubicin; Etoposide; Sargramostim; Thalidomide; Melphalan
MeSH Terms: conditions — Multiple Myeloma | interventions — Cisplatin; Cyclophosphamide; Doxorubicin; Etoposide; etoposide phosphate; Melphalan; Thalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Auto Transplant w/ High Dose Melphalan (Active Comparator): Autologous transplant with High Dose Melphalan alone
  Interventions: Drug: Melphalan
- Auto Transplant w/ Melphalan + DT Pace (Active Comparator): Melphalan plus Dexamethasone, Thalidomide, CisPlatinum, Adriamycin, Cyclophosphamide, and Etoposide
  Interventions: Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Adriamycin; Drug: Etoposide; Drug: Melphalan; Drug: Thalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Cisplatin — 20mg/m2 continuous infusion days -3 and -2.
  Other Names: Cisplatinum; cis-diamminedichloroplatinum; Platinol; Platinol-injectable (AQ)
  Arms: Auto Transplant w/ Melphalan + DT Pace
Drug: Cyclophosphamide — 800 mg/m2 continuous infusion days -3 and -2.
  Other Names: Endoxan; Cytoxan; Neosar; Procytox; Revimmune
  Arms: Auto Transplant w/ Melphalan + DT Pace
Drug: Adriamycin — 20mg/m2 continuous infusion -3 and -2.
  Other Names: hydroxydaunorubicin; Doxorubicin
  Arms: Auto Transplant w/ Melphalan + DT Pace
Drug: Etoposide — 80mg/m2 continuous infusion -3 and -2.
  Other Names: Eposin; Etopophos; Vepesid
  Arms: Auto Transplant w/ Melphalan + DT Pace
Drug: Melphalan — 200 mg/m2 IV over <20 minutes on -1 on Arm 1. 50mg/m2 IV over 20 minutes days -3 and -2 on Arm 2.
  Other Names: alkeran
Drug: Thalidomide — 200mg PO Continuing to Day +5, then hold until platelets >50 thousand (K).
  Other Names: Thalomid
  Arms: Auto Transplant w/ Melphalan + DT Pace
Drug: Dexamethasone — 40 mg po days 1 - 4 (4 days)
  Other Names: Decadron
  Arms: Auto Transplant w/ Melphalan + DT Pace

SUMMARY:
The purpose of this study is to find out if transplant with a new regimen of chemotherapy called DT PACE-Melphalan is better than transplant with Melphalan alone. DT-PACE refers to a chemotherapy regimen for multiple myeloma consisting of Dexamethasone, Thalidomide, Cisplatin or Platinol, Adriamycin or doxorubicin, Cyclophosphamide, and Etoposide. Another purpose of this study is to find out if there will be fewer side effects with the new regimen of DT PACE-Melphalan, compared to melphalan alone.

DETAILED DESCRIPTION:
To evaluate, in a randomized phase III clinical trial in previously treated multiple myeloma patients, whether angio-chemotherapy with D.T. PACE followed by tandem transplant with MEL-DTPACE Hybrid may be equivalent or superior to tandem transplant with high dose melphalan in terms of complete remission (CR)/near CR/very good partial remission (VGPR) rate and event-free and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have active multiple myeloma requiring treatment.
* Patients that have received >450 mg/m2 of prior Adriamycin therapy are eligible, however, Adriamycin will be deleted from the DT PACE regimen in these patients, unless the left ventricular ejection fraction is > 55% on Multi-gated Acquisition Scan (MUGA) or Echocardiogram (ECHO). If the patient has had > 450 mg/m2 of prior adriamycin, the LVEF must be evaluated prior to every cycle of DT PACE and it must be > 55% for patient to continue to receive adriamycin.
* All necessary baseline studies for determining eligibility must be obtained within 35 days prior to registration.
* Patients must have a performance status of 0-2 based on Southwest Oncology Group (SWOG) criteria. Patients with a poor performance status (3-4), based solely on bone pain, will be eligible.
* Patients must have a platelet count greater than or equal to 100,000/microliters. Patients with platelet count <100,000/microliters may be enrolled if it is felt to be due to extensive marrow plasmacytosis.
* Patients must have a creatinine <3 mg/dl and a creatinine clearance greater than or equal to 30 ml/minute. Patients with a creatinine clearance of 30-50 ml will only receive a 50% cisplatin dose.
* Patients must have adequate hepatic function defined as serum transaminases < 2 x Upper limit of normal (ULN) and direct bilirubin < 2.0 mg/dl.
* Patients must be able to receive full doses of DT PACE, in the opinion of the treating investigator, with some exception of: Patients that have received prior adriamycin > 450 mg/m2 and left ventricular ejection fraction (LVEF) < 55% or patients with a creatinine clearance 30 - 50 ml/minute, who will receive 50% of the cisplatin dose.
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Patients must not have significant co-morbid medical conditions or uncontrolled life threatening infection.
* Patients must not have received a prior autotransplant or allograft.
* Patients with recent (less than or equal to 6 months) myocardial infarction, unstable angina, difficult to control congestive heart failure, uncontrolled hypertension, or difficult to control cardiac arrythmias are ineligible. Ejection fraction by ECHO or must be greater than or equal to 50% and must be performed within 60 days prior to registration, unless the patient has received chemotherapy within that period of time (dexamethasone and thalidomide excluded), in which case the LVEF must be repeated.
* Patients must not have a history of chronic obstructive or chronic restrictive pulmonary disease.
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease free for at least three years.Prior malignancy is acceptable provided there has been no evidence of disease within the three-year interval.
* Pregnant or nursing women may not participate.
* Patients must not have significant co-morbid medical conditions or uncontrolled life threatening infection.
* Patients must not have a history of chronic obstructive or chronic restrictive pulmonary disease. Patients must have adequate pulmonary function studies greater than or equal to 50% of predicted on mechanical aspects (FEV1, forced vital capacity (FVC) and diffusion capacity (DLCO) greater than or equal to 50% of predicted. Patients unable to complete pulmonary function tests due to myeloma related pain or fracture must have a high resolution CT scan of the chest and must also have acceptable arterial blood gases defined as P02 greater than 70.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2001-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frits van Rhee, M.D., Ph.D., Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences/MIRT, Little Rock, Arkansas, United States

REFERENCES:
- See also: Myeloma Institute for Research & Therapy website — http://myeloma.uams.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Dose Melphalan | Mel-DT PACE
Started | 52 | 45
Completed | 2 | 8
Not Completed | 50 | 37
Not completed — Death | 6 | 3
Not completed — Physician Decision | 11 | 6
Not completed — Withdrawal by Subject | 8 | 3
Not completed — disease progression | 18 | 23
Not completed — Failure to collect | 3 | 0
Not completed — No response | 3 | 1
Not completed — Insurance issues | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Melphalan | Mel-DT PACE | Total
Number analyzed (Participants) | 52 | 45 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 24 | 51
  >=65 years | 25 | 21 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.83 (8.77) | 65.5 (8.36) | 65.14 (8.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 30 | 26 | 56

OUTCOME MEASURES:

1. Primary Outcome: Transplant With DT PACE-Melphalan Regimen of Chemotherapy vs. Transplant With Melphalan Alone.
Description: Compare a new regimen of chemotherapy called DT PACE-Melphalan (new experimental therapy) is better than transplant with Melphalan alone (standard therapy)
Time Frame: 3 years depending on start date
Population: only 2 participants in high dose (HD) melphalan group completed the study and only 8 from the Mel-DT Pace group completed the study. No analysis done.
Arm/Group | High Dose Melphalan | Mel-DT PACE
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | High Dose Melphalan | Mel-DT PACE
Serious Adverse Events (participants affected / at risk) | 6/52 | 3/45
Other Adverse Events (participants affected / at risk) | 27/52 | 24/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Melphalan (N=52) | Mel-DT PACE (N=45)
death (General disorders) | 6 (6) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Melphalan (N=52) | Mel-DT PACE (N=45)
neutropenic fever (General disorders) | 5 (5) | 4 (5)
DVT (Blood and lymphatic system disorders) | 4 (7) | 4 (5)
Diverticulitis (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
CVL infection (Infections and infestations) | 1 (1) | 1 (1)
nausea, vomiting, diarrhea & fever (Gastrointestinal disorders) | 5 (7) | 4 (5)
pneumonia (General disorders) | 3 (3) | 2 (2)
headcache, rhinitis (General disorders) | 0 (0) | 1 (1)
supraventricular tachycardia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
difficile colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
hematoma (General disorders) | 1 (1) | 1 (1)
fracture (General disorders) | 1 (1) | 1 (1)
edema (General disorders) | 0 (0) | 1 (1)
stroke (Vascular disorders) | 0 (0) | 1 (1)
hemorrhagic colitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
dehydration (General disorders) | 0 (0) | 1 (1)
drug rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
chest pain (Cardiac disorders) | 1 (1) | 0 (0)
bladder cancer (Renal and urinary disorders) | 1 (1) | 0 (0)
plasma cells in lungs (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes